CLINICAL TRIAL: NCT01835704
Title: Health-economic Evaluation of Interventional Pain Management Among Patients With Chronic Pain
Brief Title: Health-economic Evaulation of Interventional Pain Mangement
Status: Completed | Type: Observational
Sponsor: Eques Indolor AB (Other)
Responsible Party: Sponsor
Other Study IDs: SE-Dnr-2012-446-31M-2
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic pain associated to facet-joints: Patients where the pain can be localized to the facet joints.
  Interventions: Other: Radio-frequency dennervation of facet joint
- Chronic pain of other origin: Patients with pain that can not be localized to facet joints.
  Interventions: Other: Diagnostic nerve-blocks performed under direct x-ray vision

INTERVENTIONS:
Other: Radio-frequency dennervation of facet joint
  Groups: Chronic pain associated to facet-joints
Other: Diagnostic nerve-blocks performed under direct x-ray vision
  Groups: Chronic pain of other origin

SUMMARY:
To establish the cost per QALY (Quality Adjusted life Years) gained all patients that are referred to a specialized interventional pain clinic are assessed by Euroqol EQ-5D to measure the health-related quality of life at the first visit and then during the following year. Quality of life is calculated from EQ-5D by using hte TTO-validated UK-value set. With this and calculations of the cost we will be able to calculate the cost per QALY-gained which makes it possible to compare interventional pain managment to other treatments for pain patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pain of more then 6 months duration
Sampling Method: Non-Probability Sample
Enrollment: 1540 (Actual)
Dates: Start 2008-01; Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
Quality Adjusted Life gained | 1 year
  QALY is calculated from the EQ-5D value using the TTO-validated UK value set accoring to ordinary health-economic evaluations.

SECONDARY OUTCOMES:
Cost per QALY gained | 1 year
  The cost per QALY gained is calculated according to normal health-economic evaluation models.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hambraeus, MD, Principal Investigator
Locations (1):
- Smärtkliniken i Umeå, Umeå, Sweden

REFERENCES:
- [Derived] Hambraeus J, Pulkki-Brannstrom AM, Lindholm L. Cost-effectiveness of Radiofrequency Denervation for Zygapophyseal Joint Pain. Pain Physician. 2021 Dec;24(8):E1205-E1218. PMID 34793647